CLINICAL TRIAL: NCT03013894
Title: Feasibility of Confocal Laser Endomicroscopy in Bladder Cancer Diagnosis
Brief Title: Confocal Laser Endomicroscopy in the Lower Urinary Tract
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. J.J.M.C.H. de la Rosette, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2015_300
Record Dates: First submitted 2016-12-28; First posted 2017-01-09 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Bladder Neoplasm; Urothelial Carcinoma
Keywords: bladder neoplasm; urothelium carcinoma; confocal laser endomicroscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CLE images (without DNA) and histopathology (with DNA)
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: Cystoscopy and cytology, the current 'gold standard' for detection and follow-up of primary and recurrent bladder cancer have some limitations. CLE, a high resolution imaging technique, that can be used combined with endo-urological procedures, seems promising to improve diagnosis of bladder cancer. The diagnostic accuracy of cystoscopic applied confocal laser endomicroscopy (CLE) still has to be defined.

Objective: To directly correlate CLE images with histopathology, and identify and define CLE characteristics of normal urothelium, benign bladder urothelium, and bladder tumors (low-grade, high-grade and carcinoma in situ (CIS)) of the lower urinary tract.

Primary objective: to develop descriptive image interpretation criteria and a classification of CLE images of bladder tissue through a review of prospectively obtained CLE videos from bladder tissue correlated with histopathology.

Secondary objectives:

* Assessing procedure related adverse events of CLE
* Assessing technical feasibility of CLE
* To develop a CLE image atlas for urothelium of the lower urinary tract (normal, benign, low-grade or high-grade and CIS)

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational study; the investigators will establish sensitivity and specificity of CLE ex vivo and in vivo, in the diagnosis of bladder carcinoma.

Eligible patients are diagnosed with a bladder tumor at the outpatient clinic and scheduled for transurethral resection of bladder tumor (TURB). In total the investigators want to include 60 patients. Yearly approximately 70 patients are diagnosed with primary and recurrent bladder carcinoma in the Academic Medical Center (AMC) and will undergo TURB.

Their Urologist will inform patients diagnosed with a bladder tumor who will be scheduled for treatment by means of TURB about the study. Information about the study will be provided both orally and in written form.

CLE images are recorded using a probe-based system (Cellvizio 100 series, Mauna Kea Technologies, Paris, France). The probe (Cystoflex UHD-R, Mauna Kea Technologies, Paris, France) has an outer diameter of 2.8 mm, a field of view of 240 µm and has a resolution of 1 µm. Images are collected at a scan rate of 12 frames per second. Using the Cellvizio Viewer system, the investigators can observe mucosal microarchitecture with an increased field of view through mosaic post processing. This system also enables virtual staining of mucosal structures to further enhance tissue contrast.

A fluorescent contrast agent is needed to obtain CLE images. Fluorescein (fluoresceinedisodium, Fresenius Kabi, Zeist, Netherlands), a non-toxic and commonly used fluorescent dye will be administered intravesical (300-400 mL 0.1% fluorescein diluted in saline) and left indwelling for 5 minutes to stain the extracellular matrix.

The study consists of three CLE measurements, one in vivo prior to tumor resection, the second ex vivo of the resected specimen, and the last measurement is ex vivo after fixating the tumor on formaldehyde. In the case of multiple tumors, multiple CLE measurements will be done. The measurement per-operatively will add approximately 15 minutes to operating time. In the ex vivo set up, additional images will be acquired using Optical Coherence Tomography (OCT). During tumor resection, a small chip of normal urothelium will be resected additionally to act as control. Resected bladder tissue will be fixed and laminated by the pathology department, to correlate to CLE images.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Bladder tumor(s)
* Candidate for TURB
* Signed informed consent

Exclusion Criteria:

* Patients <18 years old
* Patients with known allergy for fluorescein
* Possible pregnancy or lactating women
* No signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years old with primary or recurrent bladder tumor(s), who are scheduled for TURB are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Confocal laser endomicroscopy characteristics of urothelium of the lower urinary tract | 1.5 years
  Qualitatively correlating CLE images to histopathology to define CLE characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Jean J de la Rosette, prof. dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liem EI, Freund JE, Baard J, de Bruin DM, Laguna Pes MP, Savci-Heijink CD, van Leeuwen TG, de Reijke TM, de la Rosette JJ. Confocal Laser Endomicroscopy for the Diagnosis of Urothelial Carcinoma in the Bladder and the Upper Urinary Tract: Protocols for Two Prospective Explorative Studies. JMIR Res Protoc. 2018 Feb 7;7(2):e34. doi: 10.2196/resprot.8862. PMID 29415874